CLINICAL TRIAL: NCT00966147
Title: Advanced Hemodynamic Monitoring for Goal-directed Hemodynamic Management During Radical Cystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Yuval Meroz, MD, Hadassah Medical Organization, Jerusalem, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: meroz01- HMO-CTIL
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-07

CONDITIONS: Radical Cystectomy; Perioperative Complications; Hemodynamic Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lidco group (Experimental): All patients monitored by the lidco system and treated to optimize oxygen delivery
  Interventions: Other: Increasing oxygen delivery .

INTERVENTIONS:
Other: Increasing oxygen delivery . — The target is increasing oxygen delivery above 600ml/min/mr2 by either bolus of iv colloid or a continuous infusion of dopamine, dobutamine or noradrenaline. The fluids and drug administration will be directed and monitored by the lidco system and transesophageal echocardiography.

SUMMARY:
The purpose of this study is to determine whether increasing cardiac output by a combination of intravenous fluids and inotropic drugs can reduce mortality and morbidity in radical cystectomy operations.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18yo) scheduled for elective radical cystectomy and ileal conduit formation

Exclusion Criteria:

* Creatinine level above 200 mcg/dl
* single functioning kidney
* s/p kidney transplant
* heart rhythm other than sinus
* known allergy to lithium chloride
* chronic lithium therapy
* weight below 40 kg
* mental or language problems that precludes obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-10

PRIMARY OUTCOMES:
Mortality | Hospital stay

SECONDARY OUTCOMES:
Morbidity | Hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel